CLINICAL TRIAL: NCT00988026
Title: Safety and Efficacy Comparison of Minocycline Microgranules vs Lymecycline in the Treatment of Mild to Moderate Acne. Randomized, Double Blind, Parallel and Prospective Clinical Trial for 8 Weeks
Brief Title: Safety and Efficacy Comparison of Minocycline Microgranules Versus Lymecycline in the Treatment of Mild to Moderate Acne
Acronym: MXMIN-001
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Darier (Industry)
Responsible Party: Luis Leobardo Velázquez-Arenas, Hospital "Dr. José Eleuterio González" de la Universidad Autónoma de Nuevo Léon
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MXMIN-001
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Last update posted 2009-10-01 (Estimated); Status verified 2009-09

CONDITIONS: Mild to Moderate Acne

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Minocycline 100 mg (Experimental): Minocycline
  Interventions: Drug: Minocycline vs Lymecycline
- Lymecycline 300 mg (Active Comparator): Group B: Lymecycline
  Interventions: Drug: Minocycline vs Lymecycline

INTERVENTIONS:
Drug: Minocycline vs Lymecycline — Minocycline 100 mg OD per mouth for 8 weeks. Lymecycline 300 mg OD per mouth for 8 weeks.

SUMMARY:
This is a clinical trial to compare the benefits and possible adverse events of two antibiotic treatments for mild to moderate acne. It is expected that minocycline microgranules will be more effective than lymecycline with a better adverse events profile.

ELIGIBILITY:
Inclusion Criteria:

* Both gender
* 14 to 30 years old
* Mild to moderate acne
* Face localization
* At least 20 non-inflammatory lesions OR
* At least 15 inflammatory lesions OR
* At least 30 total lesions AND
* Less than 5 nodular lesions

Exclusion Criteria:

* Patients younger than 14 or older than 30 years old
* Less than 20 non-inflammatory lesions OR
* Less than 15 inflammatory lesions OR
* Less than 30 total lesions
* Patients with severe acne
* More than 5 nodular lesions OR
* More than 50 inflammatory lesions OR
* More than 125 total lesions
* Pregnant women
* Lactating women

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 168 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-02 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Number of inflammatory and non-inflammatory acne lesions | 8 weeks

SECONDARY OUTCOMES:
Incidence of local and systemic adverse events | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Servicio de Dermatología. Hospital " Dr. José Eleuterio González" de la Universidad Autónoma de Nuevo León, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Derived] Ocampo-Candiani J, Velazquez-Arenas LL, de la Fuente-Garcia A, Trevino-Gomezharper C, Berber A. Safety and efficacy comparison of minocycline microgranules vs lymecycline in the treatment of mild to moderate acne: randomized, evaluator-blinded, parallel, and prospective clinical trial for 8 weeks. J Drugs Dermatol. 2014 Jun;13(6):671-6. PMID 24918556